CLINICAL TRIAL: NCT04146571
Title: Expanded Access Intermediate-Size Patient Population Protocol
Brief Title: Expanded Access to Ensartinib for Participants With ALK+ NSCLC
Status: Available | Type: Expanded Access
Sponsor: Xcovery Holdings, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: X396-CLI-205
Record Dates: First submitted 2019-10-28; First posted 2019-10-31 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Non-Small Cell Lung Cancer; ALK Gene Rearrangement Positive
Keywords: ensartinib; X-396; X396; anaplastic lymphoma kinase; ALK+; ALK positive; NSCLC; Non-Small Cell Lung Cancer; ALK inhibitor; carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma | interventions — ensartinib

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Ensartinib — Oral, ALK inhibitor
  Other Names: X-396; X396

SUMMARY:
This is an open-label, multicenter, intermediate-sized expanded access treatment protocol to the existing IND 111,695 for ensartinib (X-396). The treatment plan is designed to provide ensartinib to participants with anaplastic lymphoma kinase (ALK)-rearranged non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
Open-label, multi-center, intermediate-sized expanded access treatment protocol for X396-CLI-101 (Phase I/II, First-in-Human, Dose-Escalation Study of X-396 in Patients with Advanced Solid Tumors and Expansion Phase in Patients with ALK+ Non-Small Cell Lung Cancer)

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (>18 years-of-age) with advanced ALK-positive NSCLC as determined by an FDA approved test.
2. Eastern Cooperative Group (ECOG) Performance Status score of 0 or 1.
3. Informed consent must be provided by each patient.
4. Patient is not eligible or does not have access for participation in any of the other ongoing clinical trials for ensartinib.
5. Ability to swallow and retain oral medication.
6. Male and female patients must agree to abstain or to use two highly effective forms of contraception during the treatment period and for 90 days after the last dose of study medication.
7. Adequate organ system function.
8. Patients with treated CNS metastases are eligible if they are asymptomatic with respect to the CNS metastases and do not require escalating doses of systemic corticosteroids. ALK-positive patients with untreated CNS lesions may be allowed to enroll as long as the patients are asymptomatic with respect to the CNS metastases and do not require systemic corticosteroids or anticonvulsants.

Exclusion Criteria:

1. Patients currently receiving cancer therapy.
2. Use of an investigational or targeted drug within 21 days or 5 half-lives (whichever is shorter) prior to the first dose of ensartinib. A minimum of 10 days between termination of the treatment and administration of ensartinib is required. However, in the case of ALK TKIs, a 2-day window between termination of the TKI and the start of ensartinib is allowed. In addition, any drug-related toxicity should have recovered to Grade 1 or less, with the exception of alopecia.
3. Any major surgery or immunotherapy within the last 21 days (focal radiation does not require a washout period; ≥4 weeks for whole brain radiotherapy). Chemotherapy regimens with delayed toxicity within the last 4 weeks (or within the last 6 weeks for prior nitrosourea or mitomycin C). Chemotherapy regimens given continuously or on a weekly basis with limited potential for delayed toxicity within the last 2 weeks.
4. Patients with a known allergy or delayed hypersensitivity reaction to drugs chemically related to ensartinib (e.g., crizotinib) or to the active ingredient of ensartinib or to tartrazine, a dye used in the ensartinib 100 mg capsules.
5. Patients receiving CYP3A substrates with narrow therapeutic indices, strong CYP3A inhibitors, and strong CYP3A inducers.
6. Presence of active gastrointestinal (GI) disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of ensartinib.
7. Clinically significant cardiovascular disease.
8. Patients who are immunosuppressed (including known HIV infection), have a serious active infection at the time of treatment, have known hepatitis C, or have any serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
9. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
10. Have a history or the presence at baseline of pulmonary interstitial lung disease, drug-related pneumonitis, or radiation pneumonitis.
11. Females who are pregnant or breastfeeding.
12. Patient with any concurrent condition or receiving any concurrent medication that, in the investigator's opinion, would impart excessive risk associated with study participation or otherwise make it inappropriate for the patient to participate.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Stanford University, Stanford, California
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Vanderbilt University, Nashville, Tennessee
  - University of Wisconsin Carbone Cancer Ctr, Madison, Wisconsin

REFERENCES:
- [Background] Lovly CM, Heuckmann JM, de Stanchina E, Chen H, Thomas RK, Liang C, Pao W. Insights into ALK-driven cancers revealed through development of novel ALK tyrosine kinase inhibitors. Cancer Res. 2011 Jul 15;71(14):4920-31. doi: 10.1158/0008-5472.CAN-10-3879. Epub 2011 May 25. PMID 21613408
- [Result] Horn L, Infante JR, Reckamp KL, Blumenschein GR, Leal TA, Waqar SN, Gitlitz BJ, Sanborn RE, Whisenant JG, Du L, Neal JW, Gockerman JP, Dukart G, Harrow K, Liang C, Gibbons JJ, Holzhausen A, Lovly CM, Wakelee HA. Ensartinib (X-396) in ALK-Positive Non-Small Cell Lung Cancer: Results from a First-in-Human Phase I/II, Multicenter Study. Clin Cancer Res. 2018 Jun 15;24(12):2771-2779. doi: 10.1158/1078-0432.CCR-17-2398. Epub 2018 Mar 21. PMID 29563138